CLINICAL TRIAL: NCT03686241
Title: The Use of a Dynamic Compression Intramedullary Nail for Tibiotalocalcaneal Arthrodesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MedShape, Inc (Industry)
Collaborators: Saint Alphonsus Medical Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: SARMC-SPS207720
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Ankle Arthritis; Foot Arthritis
Keywords: Tibiotalocalcaneal arthrodesis; Intramedullary Nail; Sustained Compression
MeSH Terms: interventions — Arthrodesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Tibiotalocalcaneal (TTC) arthrodesis — Tibiotalocalcaneal (TTC) arthrodesis with a novel dynamic compression intramedullary nail.
Device: DynaNail — Utilization of a novel dynamic compression pseudoelastic intramedullary nail

SUMMARY:
The purpose of this study is to determine the clinical efficacy of a novel dynamic compression intramedullary nail for tibiotalocalcaneal (TTC) arthrodesis.

DETAILED DESCRIPTION:
This proposal is a collaborative effort between MedShape and the Saint Alphonsus Medical Group Foot and Ankle Clinic. This is a prospective investigation to assess the clinical outcomes of patients with a tibiotalocalcaneal arthrodesis with the Dynamic Compression Intramedullary Nail (DynaNail). We are planning on enrolling 30 patients. The assignment of the device is at the discretion of the standard of care provider, not the study investigator.

Patients with end-stage tibiotalar (ankle) and talocalcaneal (subtalar) joint arthritis from any etiology will be asked to enroll in the study. After informed consent, the patients will be asked to complete the following patient reported outcomes questionnaires (standard of care for all patients in the Foot and Ankle section): 100mm Visual Analog Scale (VAS) for pain, Short form-36 (SF-36), and the Foot and Ankle Ability Measure (FAAM). After informed consent, they will then be scheduled for surgery in a routine fashion.

The following surgical procedure is standard of care. The surgical procedure will involve both tibiotalar and talocalcaneal joint preparation through any approach (lateral, posterior, anterior with sinus tarsi). The use of supplemental bone graft is at the discretion of the treating surgeon but must be documented. The MedShape DynaNail will then be inserted according to the manufacturer's technique. The patient will be placed in a short leg splint and kept non-weight bearing. The patient will be discharged from the hospital when medically ready and follow-up in two weeks.

At two weeks, the patient will return to clinic and their splint will be removed. Non-weight bearing radiographs of the hind foot will be taken to assess the amount of travel of the compressive element. The patient will be placed in a non-weight bearing cast. The patient will then be asked to return in two weeks (4 weeks post-operatively). At this time additional non-weight bearing radiographs will be taken to assess the amount of travel of the compressive element. The patient will be asked to return at 6 weeks, 3 months, 6 months, 12 months, and 24 months after surgery. At 3 months, a CT scan will be obtained to assess healing. At each of these time-points, the same patient specific outcome questionnaires will be administered.

Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone over age 18 who has ankle and subtalar arthritis and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore the exclusion criteria will be patients who are not healthy enough to undergo surgery. Additional exclusion criteria include non-English speakers, and patients that are blind, illiterate, or are prisoners. Patients of all racial, religious, and cultural backgrounds will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ankle and Subtalar arthritis
* Failed non-operative management
* Able to understand the requirements of the study, provide written consent, and willing to comply with study protocol

Exclusion Criteria:

* Patients who do not meet the minimum age of 18 years
* Patients not healthy enough to undergo surgery
* Investigator determines that the subject is unlikely to comply with the requirements of the study
* Non-English speaker
* Blind
* Illiterate
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone age 18 and over who has ankle and subtalar arthritis and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore exclusion criteria will include patients who are not healthy enough to undergo surgery. Patients of all racial, religious, and cultural backgrounds will be included in this study. Approximately 30 patients will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Fusion | Pre-operative up to 2 years post surgery
  Fusion, as measured by radiograph and CT scan

SECONDARY OUTCOMES:
Pain - VAS | Pre-operative up to 2 years post surgery
  Change in pain as assessed by Visual Analog Scale. The scale consists of a 100 mm straight line, with patients asked to mark a dot along the line their severity level of pain, with one end representing "the worst pain imaginable" and the other end representing "no pain". "No pain" is a score of 0, with "the worst pain imaginable" representing a score of 100. The quantitative distances are grouped into the following categories: 0-4 mm = no pain, 5-44 mm = mild pain, 45-74 mm = moderate pain, and 75-100 mm = severe pain.
Function - SF-36 | Pre-operative up to 2 years post surgery
  Change in function as assessed by Short Form 36
Function - FAAM | Pre-operative up to 2 years post surgery
  Change in function as assessed by Foot and Ankle Ability Measure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Hirose, MD, Principal Investigator — Saint Alphonsus Medical Group Orthopedics Coughlin Foot and Ankle Clinic
Locations (1):
- Saint Alphonsus Medical Group Orthopedics Coughlin Foot and Ankle Clinic, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No